CLINICAL TRIAL: NCT03612193
Title: Role of the Gut Microbiome in Complex Regional Pain Syndrome
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201806182
Record Dates: First submitted 2018-07-09; First posted 2018-08-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Taxonomic and metabolomic biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Study A: Chronic >1 year
- Study A: Acute <1 year
- Study A: Household Control
- Study B: Newly Diagnosed <6 months
- Study B: Household Controls

SUMMARY:
The objective of this prospective, observational study is to determine the association between the composition of the gut microbiota and the severity and persistence of Complex Regional Pain Syndrome symptoms (Study A). The objective of Study B, a longitudinal study of microbiota biomarkers of patients with newly diagnosed CRPS is to determine if the researchers can predict which patients are more likely to recover compared to those who do not. A secondary objective of both studies is to examine cognitive flexibility in relation to outcomes (study A and B).

ELIGIBILITY:
Study A: Cross-sectional study

Inclusion criteria, cases:

* Adults over the age of 18
* Current (< 1 year duration) or former (> 1 year) diagnosis of Complex Regional Pain Syndrome by the Budapest criteria
* English as primary language
* able to consent

Inclusion criteria, controls

* Adults over age of 18
* Cohabitant of person with current or former diagnosis of CRPS

Study B: Longitudinal Study

Inclusion criteria, cases:

* Adults over the age of 18
* Recent diagnosis (<6 months) of Complex Regional Pain Syndrome by the Budapest criteria
* English as primary language
* able to consent

Inclusion criteria, controls

* Adults over age of 18
* Cohabitant of person with diagnosis of CRPS

Study A and B: Exclusion criteria, cases and controls:

* Unwilling to participate in the study
* Lives alone
* Current use of probiotics and unwilling to stop for 1 week prior to stool sample
* Pregnant or lactating
* Vegan diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pain Management Center at Washington University/Barnes-Jewish Hospital medical campus
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with taxonomic and metabolomic differences of the gut microbiome in relation to CRPS severity score | 1 visit - up to one month
  Study A
Number of participants with taxonomic and metabolomic differences of the gut microbiome in relation to recovery from CRPS | 12 months
  Study B

SECONDARY OUTCOMES:
Score results of the Stroop Color Word Test in relation to CRPS recovery | 12 months
  Study B
Logistic regression analysis for testing the association of CRPS severity score to weight in kilograms and height in meters aggregated to BMI (kilograms/meters squared) | 12 months
  Study B
Logistic regression analysis for testing the association of CRPS severity score to use of opioid analgesics | 12 months
  Study B

CONTACTS AND LOCATIONS:
Overall Officials: Lara Crock, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Chont M, Vatine JJ. Validation of proposed diagnostic criteria (the "Budapest Criteria") for Complex Regional Pain Syndrome. Pain. 2010 Aug;150(2):268-274. doi: 10.1016/j.pain.2010.04.030. Epub 2010 May 20. PMID 20493633
- [Background] Birklein F, Dimova V. Complex regional pain syndrome-up-to-date. Pain Rep. 2017 Oct 5;2(6):e624. doi: 10.1097/PR9.0000000000000624. eCollection 2017 Nov. PMID 29392238
- [Background] Birklein F, Ajit SK, Goebel A, Perez RSGM, Sommer C. Complex regional pain syndrome - phenotypic characteristics and potential biomarkers. Nat Rev Neurol. 2018 May;14(5):272-284. doi: 10.1038/nrneurol.2018.20. Epub 2018 Mar 16. PMID 29545626
- [Background] Lenz M, Uceyler N, Frettloh J, Hoffken O, Krumova EK, Lissek S, Reinersmann A, Sommer C, Stude P, Waaga-Gasser AM, Tegenthoff M, Maier C. Local cytokine changes in complex regional pain syndrome type I (CRPS I) resolve after 6 months. Pain. 2013 Oct;154(10):2142-2149. doi: 10.1016/j.pain.2013.06.039. Epub 2013 Jun 27. PMID 23811041
- [Background] Ware MA, Bennett GJ. Case report: Long-standing complex regional pain syndrome relieved by a cephalosporin antibiotic. Pain. 2014 Jul;155(7):1412-1415. doi: 10.1016/j.pain.2014.03.014. Epub 2014 Mar 22. PMID 24667741
- [Background] Weinstock LB, Myers TL, Walters AS, Schwartz OA, Younger JW, Chopra PJ, Guarino AH. Identification and Treatment of New Inflammatory Triggers for Complex Regional Pain Syndrome: Small Intestinal Bacterial Overgrowth and Obstructive Sleep Apnea. A A Case Rep. 2016 May 1;6(9):272-6. doi: 10.1213/XAA.0000000000000292. PMID 26867023
- [Background] Fung TC, Olson CA, Hsiao EY. Interactions between the microbiota, immune and nervous systems in health and disease. Nat Neurosci. 2017 Feb;20(2):145-155. doi: 10.1038/nn.4476. Epub 2017 Jan 16. PMID 28092661
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Frank DN, Robertson CE, Hamm CM, Kpadeh Z, Zhang T, Chen H, Zhu W, Sartor RB, Boedeker EC, Harpaz N, Pace NR, Li E. Disease phenotype and genotype are associated with shifts in intestinal-associated microbiota in inflammatory bowel diseases. Inflamm Bowel Dis. 2011 Jan;17(1):179-84. doi: 10.1002/ibd.21339. Epub 2010 Sep 13. PMID 20839241
- [Background] Bercik P, Denou E, Collins J, Jackson W, Lu J, Jury J, Deng Y, Blennerhassett P, Macri J, McCoy KD, Verdu EF, Collins SM. The intestinal microbiota affect central levels of brain-derived neurotropic factor and behavior in mice. Gastroenterology. 2011 Aug;141(2):599-609, 609.e1-3. doi: 10.1053/j.gastro.2011.04.052. Epub 2011 Apr 30. PMID 21683077
- [Background] Shen S, Lim G, You Z, Ding W, Huang P, Ran C, Doheny J, Caravan P, Tate S, Hu K, Kim H, McCabe M, Huang B, Xie Z, Kwon D, Chen L, Mao J. Gut microbiota is critical for the induction of chemotherapy-induced pain. Nat Neurosci. 2017 Sep;20(9):1213-1216. doi: 10.1038/nn.4606. Epub 2017 Jul 17. PMID 28714953
- [Background] Amaral FA, Sachs D, Costa VV, Fagundes CT, Cisalpino D, Cunha TM, Ferreira SH, Cunha FQ, Silva TA, Nicoli JR, Vieira LQ, Souza DG, Teixeira MM. Commensal microbiota is fundamental for the development of inflammatory pain. Proc Natl Acad Sci U S A. 2008 Feb 12;105(6):2193-7. doi: 10.1073/pnas.0711891105. Epub 2008 Feb 11. PMID 18268332
- [Background] Nayak RR, Turnbaugh PJ. Mirror, mirror on the wall: which microbiomes will help heal them all? BMC Med. 2016 May 4;14:72. doi: 10.1186/s12916-016-0622-6. PMID 27146150
- [Background] Wang F, Meng J, Zhang L, Johnson T, Chen C, Roy S. Morphine induces changes in the gut microbiome and metabolome in a morphine dependence model. Sci Rep. 2018 Feb 26;8(1):3596. doi: 10.1038/s41598-018-21915-8. PMID 29483538
- [Background] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Background] Ji RR, Chamessian A, Zhang YQ. Pain regulation by non-neuronal cells and inflammation. Science. 2016 Nov 4;354(6312):572-577. doi: 10.1126/science.aaf8924. PMID 27811267
- [Background] Powell N, Walker MM, Talley NJ. The mucosal immune system: master regulator of bidirectional gut-brain communications. Nat Rev Gastroenterol Hepatol. 2017 Mar;14(3):143-159. doi: 10.1038/nrgastro.2016.191. Epub 2017 Jan 18. PMID 28096541
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Neuman H, Debelius JW, Knight R, Koren O. Microbial endocrinology: the interplay between the microbiota and the endocrine system. FEMS Microbiol Rev. 2015 Jul;39(4):509-21. doi: 10.1093/femsre/fuu010. Epub 2015 Feb 19. PMID 25701044
- [Background] Lyte M. Microbial endocrinology in the microbiome-gut-brain axis: how bacterial production and utilization of neurochemicals influence behavior. PLoS Pathog. 2013;9(11):e1003726. doi: 10.1371/journal.ppat.1003726. Epub 2013 Nov 14. No abstract available. PMID 24244158
- [Background] Lyte M. Microbial endocrinology: Host-microbiota neuroendocrine interactions influencing brain and behavior. Gut Microbes. 2014 May-Jun;5(3):381-9. doi: 10.4161/gmic.28682. Epub 2014 Apr 1. PMID 24690573
- [Background] Nair AT, Ramachandran V, Joghee NM, Antony S, Ramalingam G. Gut Microbiota Dysfunction as Reliable Non-invasive Early Diagnostic Biomarkers in the Pathophysiology of Parkinson's Disease: A Critical Review. J Neurogastroenterol Motil. 2018 Jan 30;24(1):30-42. doi: 10.5056/jnm17105. PMID 29291606
- [Background] Nagy-Szakal D, Williams BL, Mishra N, Che X, Lee B, Bateman L, Klimas NG, Komaroff AL, Levine S, Montoya JG, Peterson DL, Ramanan D, Jain K, Eddy ML, Hornig M, Lipkin WI. Fecal metagenomic profiles in subgroups of patients with myalgic encephalomyelitis/chronic fatigue syndrome. Microbiome. 2017 Apr 26;5(1):44. doi: 10.1186/s40168-017-0261-y. PMID 28441964
- [Background] Dinsdale EA, Edwards RA, Hall D, Angly F, Breitbart M, Brulc JM, Furlan M, Desnues C, Haynes M, Li L, McDaniel L, Moran MA, Nelson KE, Nilsson C, Olson R, Paul J, Brito BR, Ruan Y, Swan BK, Stevens R, Valentine DL, Thurber RV, Wegley L, White BA, Rohwer F. Functional metagenomic profiling of nine biomes. Nature. 2008 Apr 3;452(7187):629-32. doi: 10.1038/nature06810. Epub 2008 Mar 12. PMID 18337718
- [Background] Harden RN, Maihofner C, Abousaad E, Vatine JJ, Kirsling A, Perez RSGM, Kuroda M, Brunner F, Stanton-Hicks M, Marinus J, van Hilten JJ, Mackey S, Birklein F, Schlereth T, Mailis-Gagnon A, Graciosa J, Connoly SB, Dayanim D, Massey M, Frank H, Livshitz A, Bruehl S. A prospective, multisite, international validation of the Complex Regional Pain Syndrome Severity Score. Pain. 2017 Aug;158(8):1430-1436. doi: 10.1097/j.pain.0000000000000927. PMID 28715350
- [Background] Unger MM, Spiegel J, Dillmann KU, Grundmann D, Philippeit H, Burmann J, Fassbender K, Schwiertz A, Schafer KH. Short chain fatty acids and gut microbiota differ between patients with Parkinson's disease and age-matched controls. Parkinsonism Relat Disord. 2016 Nov;32:66-72. doi: 10.1016/j.parkreldis.2016.08.019. Epub 2016 Aug 26. PMID 27591074
- [Derived] Crock LW, Rodgers R, Huck NA, Schriefer LA, Lawrence D, Wang L, Muwanga GPB, Tawfik VL, Baldridge MT. Chronic pain and complex regional pain syndrome are associated with alterations to the intestinal microbiota in both humans and mice. An observational cross-sectional study. Neurobiol Pain. 2024 Nov 25;16:100173. doi: 10.1016/j.ynpai.2024.100173. eCollection 2024 Jul-Dec. PMID 39670171